CLINICAL TRIAL: NCT04154514
Title: A Wearable for Post-stroke Rehabilitative Multi-muscle Stimulation Inspired by the Natural Organization of Neuromuscular Control
Brief Title: A Potential Wearable for Post-stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: The Hong Kong Polytechnic University (Other); City University of Hong Kong (Other); Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Cheung Chi Kwan Vincent, Assistant Professor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREC_RIF_PROTOCOL version 01
Record Dates: First submitted 2019-10-10; First posted 2019-11-06 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Chronic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delivering FES to stroke survivors (Experimental): In stroke survivors, normal and abnormal muscle synergies will also be determined from their walk EMGs. Our proposed FES intervention involves delivering stimulations to muscles with waveforms generated from the activations of all the normal synergies not observed in each stroke survivor. We are going to employ the wearable to deliver personalized muscle-synergy-based FES stimulations to multiple groups of leg muscles on the stroke-affected side of elderly chronic stroke survivors as they walk on a treadmill/overground for gait rehabilitation. We hypothesized that the subject will essentially be walking with his/her abnormal muscle pattern superimposed with the artificially introduced "normal" muscle pattern coming from FES.
  Interventions: Device: A functional electrical stimulation device for post-stroke rehabilitation
- Delivery no current FES to stroke survivors (Sham group) (Experimental): In stroke survivors, normal and abnormal muscle synergies will also be determined from their walk EMGs. Our proposed FES intervention involves delivering stimulations to muscles with waveforms generated from the activations of all the normal synergies not observed in each stroke survivor. Additionally, we are going to introduce a sham group. We are going to employ the wearable to multiple groups of leg muscles on the stroke-affected side of elderly chronic stroke survivors without any stimulation as they walk on a treadmill or overground for gait rehabilitation. The purpose of the sham group is to empirically validate the effectiveness of the FES wearable.
  Interventions: Device: A functional electrical stimulation device for post-stroke rehabilitation

INTERVENTIONS:
Device: A functional electrical stimulation device for post-stroke rehabilitation — Most of the FDA-approved commercial FES devices deliver therapy that targets specific kinematic impairment in the step cycle (e.g., foot drop). Our device will be unique in that it can stimulate many muscles around multiple joints for a more comprehensive and naturalistic restoration of lower-limb motor functions.

SUMMARY:
Participants are seeking to unleash the full therapeutic potential of a newly developed, customizable and potentially commericializable 10-channel Functional Electrical Stimulation (FES) to rehabilitate the gait of chronic stroke survivors. Each subject will undergo 18-sessions (~1 month) FES training. Participants will utilize the theory of muscle synergies from motor neurosciences, which are defined as neural modules of motor control that coordinate the spatiotemporal activation patterns of multiple muscles, to guide our personal selections of muscles for FES. It is hypothesized that chronic stroke survivors will learn from FES stimulations, over several daily sessions, both by suppressing the original abnormal muscle synergies and by employing the normal muscle synergies as specified in the FES. It is also expected that the walk synergies of the paretic side of chronic stroke survivors should be more similar to healthy muscle synergies at the two post-training time points than before training.

DETAILED DESCRIPTION:
Stroke is one of the leading causes of long-term adult disability worldwide. The impaired ability to walk post-stroke severely limits mobility and quality of life. Many recently-developed assistive technologies for gait rehabilitation are at present only marginally better at best than traditional therapies in their efficacies. There is an urgent need of novel, clinically viable, and effective gait rehabilitative strategies that can provide even better functional outcome for stroke survivors with diverse presentations.

Among the many new post-stroke interventions, functional electrical stimulation (FES) of muscles remains attractive. FES is a neural-rehabilitative technology that communicates control signals from an external device to the neuromuscular system. There is increasing recognition that rehabilitation paradigms should promote restitution of the patient's muscle coordination towards the normal pattern during training, and FES can achieve this goal when stimulations are applied to the set of muscles whose natural coordination is impaired. For this reason, FES is a very promising interventional strategy. Existing FES paradigms, however, have yielded ambiguous results in previous clinical trials, especially those for chronic survivors, likely because either stimulations were applied only to single or a few muscles, or the stimulation pattern did not mimic the natural muscle coordination pattern during gait. A multi-muscle FES, when applied to a larger functional set of muscles and driven by their natural coordination pattern, can guide muscle activations towards the normal pattern through neuroplasticity, thus restore impairment at the level of muscle-activation deficit.

The first aim of our project is to utilize a 8-channel FES wearable for delivering multi-muscle FES to muscles in the lower-limb muscles. Participants will attempt to rehabilitate the gait of chronic stroke survivors over 12 training sessions by delivering stimulations to multiple muscles, in their natural coordination pattern, using our wearable. As such, participants will utilize the theory of muscle synergy from motor neuroscience to guide our personalizable selections of muscles for FES. Muscle synergies are hypothesized neural modules of motor control that coordinate the spatiotemporal activation patterns of multiple muscles. Our customizable FES pattern for each stroke survivor will be constructed based on the normal muscle synergies that are absent in the stroke survivor's muscle pattern during walking. Since muscle synergies represent the natural motor-control units used by the nervous system, reinforcement of their activations through FES should lead to restoration of normal neuromuscular coordination, thus more natural post-training gait.

Our second aim is to evaluate the effectiveness of our FES paradigm by assessing the walk-muscle synergies in the paretic and non-paretic legs of the trained stroke survivors, before, after, and 1 month following our intervention. In doing so, participants hope to explore whether lower-limb muscle synergy can be a physiologically-based marker of motor impairment for stroke survivors.

If our muscle-synergy-based multi-muscle FES is indeed efficacious, our strategy will help many disabled chronic stroke survivors to regain mobility, thus living with a much higher quality of life in the decades to come. The clinical and societal impact of our research will be huge.

ELIGIBILITY:
Inclusion Criteria:

1. Right-handed elderly chronic stroke survivors; age ≥40; ≥6 months post-stroke
2. Unilateral ischemic brain lesions
3. Participants should be able to walk continuously for ≥15 min. with or without assistive aid

Exclusion Criteria:

1. Cannot comprehend and follow instructions, or with a score <21 on the mini-mental state exam;
2. Have cardiac pacemaker;
3. Have skin lesions at the locations where FES or EMG electrodes may be attached;
4. Have major depression;
5. Present with severe neglect
6. Patients with type i and ii diabetes

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Surface electromyographic signals from up to 14 muscles on the paretic and non-paretic side during gait. | The assessment will be performed at baseline
  To assess the muscle synergies, surface EMGs will be recorded from 14 muscles (tibialis anterior (TA), medical gastrocnemius (MG), soleus (SOL), vastus medialis (VM), rectus femoris (RF), hamstrings (HAM), adductor longus (AL), gluteus maximus (GM) lateral gastrocnemius (LG), vastus lateralis (VL), tensor fasciae latae (TFL), erector spinae (ES), external oblique (EO), and latissimus dorsi (LatDor)), using a wireless EMG system (Delsys; 2000 Hz). All electrodes will be securely attached to skin surface using double-sided and medical tapes.
Surface electromyographic signals from up to 14 muscles on the paretic and non-paretic side during gait. | The assessment will be performed at 5.5 weeks
  To assess the muscle synergies, surface EMGs will be recorded from 14 muscles (tibialis anterior (TA), medical gastrocnemius (MG), soleus (SOL), vastus medialis (VM), rectus femoris (RF), hamstrings (HAM), adductor longus (AL), gluteus maximus (GM) lateral gastrocnemius (LG), vastus lateralis (VL), tensor fasciae latae (TFL), erector spinae (ES), external oblique (EO), and latissimus dorsi (LatDor)), using a wireless EMG system (Delsys; 2000 Hz). All electrodes will be securely attached to skin surface using double-sided and medical tapes.
Surface electromyographic signals from up to 14 muscles on the paretic and non-paretic side during gait. | The assessment will be performed at 2.5 weeks
  To assess the muscle synergies, surface EMGs will be recorded from 14 muscles (tibialis anterior (TA), medical gastrocnemius (MG), soleus (SOL), vastus medialis (VM), rectus femoris (RF), hamstrings (HAM), adductor longus (AL), gluteus maximus (GM) lateral gastrocnemius (LG), vastus lateralis (VL), tensor fasciae latae (TFL), erector spinae (ES), external oblique (EO), and latissimus dorsi (LatDor)), using a wireless EMG system (Delsys; 2000 Hz). All electrodes will be securely attached to skin surface using double-sided and medical tapes.

SECONDARY OUTCOMES:
Gait kinemetics | The assessment will be performed at baseline
  During FES sessions, kinematic measurements will be provided by the wearable's IMUs. During sessions of motor-impairment assessments, we will capture more precise kinematics using a 10-camera motion capture system (VICON; 200 Hz). This system tracks the 3D positions of 40 markers placed on the legs and torso, and is equipped with suitable models for reconstructing bilateral angles of the hip, knee and ankle.
Gait kinemetics | The assessment will be performed at 5.5 weeks
  During FES sessions, kinematic measurements will be provided by the wearable's IMUs. During sessions of motor-impairment assessments, we will capture more precise kinematics using a 10-camera motion capture system (VICON; 200 Hz). This system tracks the 3D positions of 40 markers placed on the legs and torso, and is equipped with suitable models for reconstructing bilateral angles of the hip, knee and ankle.
Gait kinemetics | The assessment will be performed at 2.5 weeks
  During FES sessions, kinematic measurements will be provided by the wearable's IMUs. During sessions of motor-impairment assessments, we will capture more precise kinematics using a 10-camera motion capture system (VICON; 200 Hz). This system tracks the 3D positions of 40 markers placed on the legs and torso, and is equipped with suitable models for reconstructing bilateral angles of the hip, knee and ankle.
Gait kinemetics | The assessment will be performed at 4 weeks
  During FES sessions, kinematic measurements will be provided by the wearable's IMUs. During sessions of motor-impairment assessments, we will capture more precise kinematics using a 10-camera motion capture system (VICON; 200 Hz). This system tracks the 3D positions of 40 markers placed on the legs and torso, and is equipped with suitable models for reconstructing bilateral angles of the hip, knee and ankle.
Fugl-Meyer assessment score (lower-limb) | The assessment will be performed at baseline
  Lower-limb motor function assessment
Fugl-Meyer assessment score (lower-limb) | The assessment will be performed at 5.5 weeks
  Lower-limb motor function assessment
Fugl-Meyer assessment score (lower-limb) | The assessment will be performed at 2.5 weeks
  Lower-limb motor function assessment
Fugl-Meyer assessment score (lower-limb) | The assessment will be performed at 4 weeks
  Lower-limb motor function assessment
Mini-BEStest | The assessment will be performed at baseline
  Balance test
Mini-BEStest | The assessment will be performed at 5.5 weeks
  Balance test
Mini-BEStest | The assessment will be performed at 2.5 weeks
  Balance test
Mini-BEStest | The assessment will be performed at 4 weeks
  Balance test

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Perry J, Garrett M, Gronley JK, Mulroy SJ. Classification of walking handicap in the stroke population. Stroke. 1995 Jun;26(6):982-9. doi: 10.1161/01.str.26.6.982. PMID 7762050
- [Background] Krasovsky T, Levin MF. Review: toward a better understanding of coordination in healthy and poststroke gait. Neurorehabil Neural Repair. 2010 Mar-Apr;24(3):213-24. doi: 10.1177/1545968309348509. Epub 2009 Oct 12. PMID 19822722
- [Background] Kollen BJ, Lennon S, Lyons B, Wheatley-Smith L, Scheper M, Buurke JH, Halfens J, Geurts AC, Kwakkel G. The effectiveness of the Bobath concept in stroke rehabilitation: what is the evidence? Stroke. 2009 Apr;40(4):e89-97. doi: 10.1161/STROKEAHA.108.533828. Epub 2009 Jan 29. PMID 19182079
- [Background] Cho JE, Yoo JS, Kim KE, Cho ST, Jang WS, Cho KH, Lee WH. Systematic Review of Appropriate Robotic Intervention for Gait Function in Subacute Stroke Patients. Biomed Res Int. 2018 Feb 6;2018:4085298. doi: 10.1155/2018/4085298. eCollection 2018. PMID 29546057
- [Background] Peckham PH, Knutson JS. Functional electrical stimulation for neuromuscular applications. Annu Rev Biomed Eng. 2005;7:327-60. doi: 10.1146/annurev.bioeng.6.040803.140103. PMID 16004574
- [Background] Sheffler LR, Chae J. Neuromuscular electrical stimulation in neurorehabilitation. Muscle Nerve. 2007 May;35(5):562-90. doi: 10.1002/mus.20758. PMID 17299744
- [Background] LIBERSON WT, HOLMQUEST HJ, SCOT D, DOW M. Functional electrotherapy: stimulation of the peroneal nerve synchronized with the swing phase of the gait of hemiplegic patients. Arch Phys Med Rehabil. 1961 Feb;42:101-5. No abstract available. PMID 13761879
- [Background] Heller BW, Clarke AJ, Good TR, Healey TJ, Nair S, Pratt EJ, Reeves ML, van der Meulen JM, Barker AT. Automated setup of functional electrical stimulation for drop foot using a novel 64 channel prototype stimulator and electrode array: results from a gait-lab based study. Med Eng Phys. 2013 Jan;35(1):74-81. doi: 10.1016/j.medengphy.2012.03.012. Epub 2012 May 4. PMID 22559959
- [Background] Springer S, Vatine JJ, Wolf A, Laufer Y. The effects of dual-channel functional electrical stimulation on stance phase sagittal kinematics in patients with hemiparesis. J Electromyogr Kinesiol. 2013 Apr;23(2):476-82. doi: 10.1016/j.jelekin.2012.10.017. Epub 2012 Dec 8. PMID 23231828
- [Background] You G, Liang H, Yan T. Functional electrical stimulation early after stroke improves lower limb motor function and ability in activities of daily living. NeuroRehabilitation. 2014;35(3):381-9. doi: 10.3233/NRE-141129. PMID 25227538
- [Background] Daly JJ, Roenigk K, Holcomb J, Rogers JM, Butler K, Gansen J, McCabe J, Fredrickson E, Marsolais EB, Ruff RL. A randomized controlled trial of functional neuromuscular stimulation in chronic stroke subjects. Stroke. 2006 Jan;37(1):172-8. doi: 10.1161/01.STR.0000195129.95220.77. Epub 2005 Dec 1. PMID 16322492
- [Background] Alon G. Use of neuromuscular electrical stimulation in neureorehabilitation: a challenge to all. J Rehabil Res Dev. 2003 Nov-Dec;40(6):ix-xii. doi: 10.1682/jrrd.2003.11.0009. No abstract available. PMID 15077655
- [Background] Alon G, Levitt AF, McCarthy PA. Functional electrical stimulation enhancement of upper extremity functional recovery during stroke rehabilitation: a pilot study. Neurorehabil Neural Repair. 2007 May-Jun;21(3):207-15. doi: 10.1177/1545968306297871. Epub 2007 Mar 16. PMID 17369518
- [Background] Cauraugh JH, Kim SB. Chronic stroke motor recovery: duration of active neuromuscular stimulation. J Neurol Sci. 2003 Nov 15;215(1-2):13-9. doi: 10.1016/s0022-510x(03)00169-2. PMID 14568122
- [Background] Saltiel P, Wyler-Duda K, D'Avella A, Tresch MC, Bizzi E. Muscle synergies encoded within the spinal cord: evidence from focal intraspinal NMDA iontophoresis in the frog. J Neurophysiol. 2001 Feb;85(2):605-19. doi: 10.1152/jn.2001.85.2.605. PMID 11160497
- [Background] Ivanenko YP, Poppele RE, Lacquaniti F. Five basic muscle activation patterns account for muscle activity during human locomotion. J Physiol. 2004 Apr 1;556(Pt 1):267-82. doi: 10.1113/jphysiol.2003.057174. Epub 2004 Jan 14. PMID 14724214
- [Background] d'Avella A, Saltiel P, Bizzi E. Combinations of muscle synergies in the construction of a natural motor behavior. Nat Neurosci. 2003 Mar;6(3):300-8. doi: 10.1038/nn1010. PMID 12563264
- [Background] Bernstein N (1967) The co-ordination and regulation of movements. Oxf. PergamoPress.
- [Background] Ting LH, Chiel HJ, Trumbower RD, Allen JL, McKay JL, Hackney ME, Kesar TM. Neuromechanical principles underlying movement modularity and their implications for rehabilitation. Neuron. 2015 Apr 8;86(1):38-54. doi: 10.1016/j.neuron.2015.02.042. PMID 25856485
- [Background] McMorland AJ, Runnalls KD, Byblow WD. A neuroanatomical framework for upper limb synergies after stroke. Front Hum Neurosci. 2015 Feb 16;9:82. doi: 10.3389/fnhum.2015.00082. eCollection 2015. PMID 25762917
- [Background] Tresch MC, Cheung VC, d'Avella A. Matrix factorization algorithms for the identification of muscle synergies: evaluation on simulated and experimental data sets. J Neurophysiol. 2006 Apr;95(4):2199-212. doi: 10.1152/jn.00222.2005. Epub 2006 Jan 4. PMID 16394079
- [Background] Brunnström S (1970) Movement therapy in hemiplegia: a neurophysiological approach. Medical Dept., Harper & Row.
- [Background] Saltiel P, Wyler-Duda K, d'Avella A, Ajemian RJ, Bizzi E. Localization and connectivity in spinal interneuronal networks: the adduction-caudal extension-flexion rhythm in the frog. J Neurophysiol. 2005 Sep;94(3):2120-38. doi: 10.1152/jn.00117.2005. Epub 2005 May 31. PMID 15928065
- [Background] Saltiel P, d'Avella A, Wyler-Duda K, Bizzi E. Synergy temporal sequences and topography in the spinal cord: evidence for a traveling wave in frog locomotion. Brain Struct Funct. 2016 Nov;221(8):3869-3890. doi: 10.1007/s00429-015-1133-5. Epub 2015 Oct 26. PMID 26501407
- [Background] Levine AJ, Hinckley CA, Hilde KL, Driscoll SP, Poon TH, Montgomery JM, Pfaff SL. Identification of a cellular node for motor control pathways. Nat Neurosci. 2014 Apr;17(4):586-93. doi: 10.1038/nn.3675. Epub 2014 Mar 9. PMID 24609464
- [Background] Cheung VC, d'Avella A, Bizzi E. Adjustments of motor pattern for load compensation via modulated activations of muscle synergies during natural behaviors. J Neurophysiol. 2009 Mar;101(3):1235-57. doi: 10.1152/jn.01387.2007. Epub 2008 Dec 17. PMID 19091930
- [Background] Cheung VC, d'Avella A, Tresch MC, Bizzi E. Central and sensory contributions to the activation and organization of muscle synergies during natural motor behaviors. J Neurosci. 2005 Jul 6;25(27):6419-34. doi: 10.1523/JNEUROSCI.4904-04.2005. PMID 16000633
- [Background] Caggiano V, Cheung VC, Bizzi E. An Optogenetic Demonstration of Motor Modularity in the Mammalian Spinal Cord. Sci Rep. 2016 Oct 13;6:35185. doi: 10.1038/srep35185. PMID 27734925
- [Background] Bizzi E, Mussa-Ivaldi FA, Giszter S. Computations underlying the execution of movement: a biological perspective. Science. 1991 Jul 19;253(5017):287-91. doi: 10.1126/science.1857964.
- [Background] Takei T, Confais J, Tomatsu S, Oya T, Seki K. Neural basis for hand muscle synergies in the primate spinal cord. Proc Natl Acad Sci U S A. 2017 Aug 8;114(32):8643-8648. doi: 10.1073/pnas.1704328114. Epub 2017 Jul 24. PMID 28739958
- [Background] Zhuang C, Marquez J, Qu H, He X, Lan N (2015) A neuromuscular electrical stimulation strategy based on muscle synergy for stroke rehabilitation. 2015:816-819.
- [Background] He X, Du YF, Lan N. Evaluation of feedforward and feedback contributions to hand stiffness and variability in multijoint arm control. IEEE Trans Neural Syst Rehabil Eng. 2013 Jul;21(4):634-47. doi: 10.1109/TNSRE.2012.2234479. Epub 2012 Dec 20. PMID 23268385
- [Background] Niu C, Zhuang C, Bao Y, Li S, Lan N, Xie Q (2017)
- [Background] Niu C (2018) Effectiveness of Short-Term Training with a Synergy-Based FES Paradigm on Motor Function Recovery Post Stroke, in 12th International Society of Physical and Rehabilitation Medicine World Congress (Paris, France).
- [Background] Ferrante S, Chia Bejarano N, Ambrosini E, Nardone A, Turcato AM, Monticone M, Ferrigno G, Pedrocchi A. A Personalized Multi-Channel FES Controller Based on Muscle Synergies to Support Gait Rehabilitation after Stroke. Front Neurosci. 2016 Sep 16;10:425. doi: 10.3389/fnins.2016.00425. eCollection 2016. PMID 27695397
- [Background] Barreca S, Wolf SL, Fasoli S, Bohannon R. Treatment interventions for the paretic upper limb of stroke survivors: a critical review. Neurorehabil Neural Repair. 2003 Dec;17(4):220-6. doi: 10.1177/0888439003259415. PMID 14677218
- [Background] Bernhardt J, Borschmann K, Boyd L, Carmichael ST, Corbett D, Cramer SC, Hoffmann T, Kwakkel G, Savitz S, Saposnik G, Walker M, Ward N. Moving Rehabilitation Research Forward: Developing Consensus Statements for Rehabilitation and Recovery Research. Neurorehabil Neural Repair. 2017 Aug;31(8):694-698. doi: 10.1177/1545968317724290. PMID 28803534
- [Background] Fugl-Meyer AR, Jaasko L, Leyman I, Olsson S, Steglind S. The post-stroke hemiplegic patient. 1. a method for evaluation of physical performance. Scand J Rehabil Med. 1975;7(1):13-31. PMID 1135616
- [Background] Dipietro L, Krebs HI, Fasoli SE, Volpe BT, Stein J, Bever C, Hogan N. Changing motor synergies in chronic stroke. J Neurophysiol. 2007 Aug;98(2):757-68. doi: 10.1152/jn.01295.2006. Epub 2007 Jun 6. PMID 17553941
- [Background] Bowden MG, Clark DJ, Kautz SA. Evaluation of abnormal synergy patterns poststroke: relationship of the Fugl-Meyer Assessment to hemiparetic locomotion. Neurorehabil Neural Repair. 2010 May;24(4):328-37. doi: 10.1177/1545968309343215. Epub 2009 Sep 30. PMID 19794132
- [Background] Gladstone DJ, Danells CJ, Black SE. The fugl-meyer assessment of motor recovery after stroke: a critical review of its measurement properties. Neurorehabil Neural Repair. 2002 Sep;16(3):232-40. doi: 10.1177/154596802401105171. PMID 12234086
- [Background] Levin MF, Kleim JA, Wolf SL. What do motor "recovery" and "compensation" mean in patients following stroke? Neurorehabil Neural Repair. 2009 May;23(4):313-9. doi: 10.1177/1545968308328727. Epub 2008 Dec 31. PMID 19118128
- [Background] Safavynia SA, Torres-Oviedo G, Ting LH. Muscle Synergies: Implications for Clinical Evaluation and Rehabilitation of Movement. Top Spinal Cord Inj Rehabil. 2011 Summer;17(1):16-24. doi: 10.1310/sci1701-16. PMID 21796239
- [Background] Stinear CM, Barber PA, Smale PR, Coxon JP, Fleming MK, Byblow WD. Functional potential in chronic stroke patients depends on corticospinal tract integrity. Brain. 2007 Jan;130(Pt 1):170-80. doi: 10.1093/brain/awl333. PMID 17148468
- [Background] Kim B, Winstein C. Can Neurological Biomarkers of Brain Impairment Be Used to Predict Poststroke Motor Recovery? A Systematic Review. Neurorehabil Neural Repair. 2017 Jan;31(1):3-24. doi: 10.1177/1545968316662708. Epub 2016 Aug 8. PMID 27503908
- [Background] Cheung VC, Piron L, Agostini M, Silvoni S, Turolla A, Bizzi E. Stability of muscle synergies for voluntary actions after cortical stroke in humans. Proc Natl Acad Sci U S A. 2009 Nov 17;106(46):19563-8. doi: 10.1073/pnas.0910114106. Epub 2009 Oct 30. PMID 19880747
- [Background] Roh J, Rymer WZ, Perreault EJ, Yoo SB, Beer RF. Alterations in upper limb muscle synergy structure in chronic stroke survivors. J Neurophysiol. 2013 Feb;109(3):768-81. doi: 10.1152/jn.00670.2012. Epub 2012 Nov 14. PMID 23155178
- [Background] Li S, Zhuang C, Niu CM, Bao Y, Xie Q, Lan N. Evaluation of Functional Correlation of Task-Specific Muscle Synergies with Motor Performance in Patients Poststroke. Front Neurol. 2017 Jul 19;8:337. doi: 10.3389/fneur.2017.00337. eCollection 2017. PMID 28785238
- [Background] Clark DJ, Ting LH, Zajac FE, Neptune RR, Kautz SA. Merging of healthy motor modules predicts reduced locomotor performance and muscle coordination complexity post-stroke. J Neurophysiol. 2010 Feb;103(2):844-57. doi: 10.1152/jn.00825.2009. Epub 2009 Dec 9. PMID 20007501
- [Background] Barroso FO, Torricelli D, Molina-Rueda F, Alguacil-Diego IM, Cano-de-la-Cuerda R, Santos C, Moreno JC, Miangolarra-Page JC, Pons JL. Combining muscle synergies and biomechanical analysis to assess gait in stroke patients. J Biomech. 2017 Oct 3;63:98-103. doi: 10.1016/j.jbiomech.2017.08.006. Epub 2017 Aug 20. PMID 28882330
- [Background] Routson RL, Clark DJ, Bowden MG, Kautz SA, Neptune RR. The influence of locomotor rehabilitation on module quality and post-stroke hemiparetic walking performance. Gait Posture. 2013 Jul;38(3):511-7. doi: 10.1016/j.gaitpost.2013.01.020. Epub 2013 Mar 13. PMID 23489952
- [Background] Hashiguchi Y, Ohata K, Kitatani R, Yamakami N, Sakuma K, Osako S, Aga Y, Watanabe A, Yamada S. Merging and Fractionation of Muscle Synergy Indicate the Recovery Process in Patients with Hemiplegia: The First Study of Patients after Subacute Stroke. Neural Plast. 2016;2016:5282957. doi: 10.1155/2016/5282957. Epub 2016 Dec 19. PMID 28090358
- [Background] Lee DD, Seung HS. Learning the parts of objects by non-negative matrix factorization. Nature. 1999 Oct 21;401(6755):788-91. doi: 10.1038/44565. PMID 10548103
- [Background] Cerina L, Cancian P, Franco G, Santambrogio M (2017) A hardware acceleration for surface EMG non-negative matrix factorization. IEEE Int Parallel & Distributed Processing Symposium Workshops 2017: 168-74.
- [Background] Santuz A, Ekizos A, Janshen L, Baltzopoulos V, Arampatzis A. On the Methodological Implications of Extracting Muscle Synergies from Human Locomotion. Int J Neural Syst. 2017 Aug;27(5):1750007. doi: 10.1142/S0129065717500071. Epub 2016 Sep 23. PMID 27873551
- [Background] Devarajan K, Cheung VC. On nonnegative matrix factorization algorithms for signal-dependent noise with application to electromyography data. Neural Comput. 2014 Jun;26(6):1128-68. doi: 10.1162/NECO_a_00576. Epub 2014 Mar 31. PMID 24684448
- [Background] Ivanenko YP, Poppele RE, Lacquaniti F. Spinal cord maps of spatiotemporal alpha-motoneuron activation in humans walking at different speeds. J Neurophysiol. 2006 Feb;95(2):602-18. doi: 10.1152/jn.00767.2005. Epub 2005 Nov 9. PMID 16282202
- [Background] Bohannon RW. Comfortable and maximum walking speed of adults aged 20-79 years: reference values and determinants. Age Ageing. 1997 Jan;26(1):15-9. doi: 10.1093/ageing/26.1.15. PMID 9143432
- [Background] Cheung VC, Turolla A, Agostini M, Silvoni S, Bennis C, Kasi P, Paganoni S, Bonato P, Bizzi E. Muscle synergy patterns as physiological markers of motor cortical damage. Proc Natl Acad Sci U S A. 2012 Sep 4;109(36):14652-6. doi: 10.1073/pnas.1212056109. Epub 2012 Aug 20. PMID 22908288
- [Background] Dominici N, Ivanenko YP, Cappellini G, d'Avella A, Mondi V, Cicchese M, Fabiano A, Silei T, Di Paolo A, Giannini C, Poppele RE, Lacquaniti F. Locomotor primitives in newborn babies and their development. Science. 2011 Nov 18;334(6058):997-9. doi: 10.1126/science.1210617. PMID 22096202
- [Background] Bizzi E, Cheung VC. The neural origin of muscle synergies. Front Comput Neurosci. 2013 Apr 29;7:51. doi: 10.3389/fncom.2013.00051. eCollection 2013. PMID 23641212